CLINICAL TRIAL: NCT06224075
Title: Task-specific Training for Patients With Acute Exacerbation of COPD
Acronym: COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Chair of Physiotherapy, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DF0101UG
Record Dates: First submitted 2024-01-12; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task-specific training (Experimental)
  Interventions: Behavioral: Task-specific training; Other: Usual care
- Usual care (Other)
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Task-specific training — Participants in the intervention group will receive the treatment established for the control group and nursing care based on task-specific training. The intervention was designed with the aim of improving inhaler management in COPD patients. The content of the tasks will be adapted to the different types of devices present in the patient's therapeutic regimen, mainly pressurized cartridge and dry powder devices.
  In order to carry out the intervention, several tasks related to education, assessment and/or training will be established with the aim of improving the ability to use the prescribed inhalers. The tasks have been classified into 3 blocks: technique execution, device cleaning and medication administration.
  Arms: Task-specific training
Other: Usual care — All patients will receive standard treatment during their hospital stay (medical and pharmacological care). This treatment will include steroids, antibiotics, inhaled bronchodilators and oxygen therapy. In addition, during hospitalization they may receive diuretics, anticoagulants and cardiovascular treatments if necessary.

SUMMARY:
Patients with Chronic Obstructive Pulmonary Disease (COPD) experience a progressive deterioration in their quality of life. Task-specific training is a type of approach focused on chronic patients that allows the acquisition of new skills or improvement of lost skills. The overall objective of this project is to evaluate the effectiveness of a task-specific training program during hospitalization of patients with acute exacerbation of COPD. A randomized clinical trial will be conducted in patients hospitalized for COPD. Participants after signing informed consent will be randomized between the control group (standard treatment) and the intervention group (task-specific training program in addition to standard treatment). The task-specific training program is a multidisciplinary program divided into three blocks where specific tasks will be performed on symptom education, education of activities of daily living and improvement of physical capacity with the aim of reinforcing skills necessary for the self-management of COPD patients in the short, medium and long term.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for acute exacerbation of COPD.
* Over 18 years of age.
* Who wish to participate in the study.
* Who sign the informed consent form.

Exclusion Criteria:

* Patients with inability to provide informed consent.
* Presence of psychiatric or cognitive disorders, organ failure, cancer and/or inability to cooperate.
* Patients who had experienced exacerbation of COPD in the previous month were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Modified Borg Scale | Baseline, hospital discharge, 1 month, 3 months and 6 months
  the perceived dyspnoea is measure with the Borg Scale. This scale range from 0-10 where higher value indicate worse state, more dyspnoea.
COPD Assessment Test (CAT) | Baseline, hospital discharge, 1 month, 3 months and 6 months
  It consists of eight questions covering cough, phlegm, chest tightness, breathlessness, activity limitations at home, confidence leaving home, sleep and energy. The items are graded from 0 to 5, giving a total score range from 0 to 40, where lower scores indicate fewer symptoms and a better quality of life.
EuroQol-5D (EQ-5D) | Baseline, hospital discharge, 1 month, 3 months and 6 months
  Changes in quality of life were measured using the Euroqol 5dimensions which comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. It also includes a visual analogue scale to report the health status from 0 to 100. Higher score indicate higher quality of life. Better.
Chronic Obstructive Pulmonary Disease Knowledge Questionnaire (COPD-Q) | Baseline, 1 months and 6 months
  Evaluated at baseline by Chronic Obstructive Pulmonary Disease Questionnaire (COPD-Q). COPD knowledge was evaluated using the Chronic Obstructive Pulmonary Disease Knowledge Questionnaire (COPD-Q; Maples, Franks, Ray, Stevens, & Wallace, 2010). The COPD-Q is a valid, readable, and reliable 13-item (each one score 0 to 3) self-administered true/false questionnaire assessing COPD knowledge in patients with low health literacy skills. A higher punctuation indicates better results.
Test of Adherence to Inhalers (TAI) | Baseline, hospital discharge, 1 month, 3 months and 6 months
  This questionnaire has two forms, the first type being a 10-item to identify the patient's adherence status to inhalers. There are 2 other questions to check the degree of compliance. The 10-item form is scored from 1 (the poorest) to 5(the best) for each item, and the total score of the questionnaire ranges from 10 to 50 (a score of 45 or less indicates poor adherence, 46 to 49 is intermediate adherence, and 50 indicates good adherence

SECONDARY OUTCOMES:
Forced expiratory volume in the first second (FEV1) | Baseline and hospital discharge
  Changes from baseline to postintervention in FEV1vas evaluated by a spirometer.
Pressure expiratory force (PEF) | Baseline and hospital discharge
  Changes from baseline to post-intervention in PEF were assessed using a peak flow
Pressure inspiratory force (PIF) | Baseline and hospital discharge
  Changes from baseline to post-intervention in PEF were assessed using a check-dial.
Technique of the inhaler | Baseline and hospital discharge
  The evaluation of the technique of the inhalers was carried out by means of a checklist composed of 5 items. Checked those points that were done correctly obtaining 5 points if the technique that was done correctly.
Postural evaluation | Baseline and hospital discharge
  Using photometry with anatomical landmarks established in this population
Patient activation measure (PAM) | Baseline, 1 month and 6 months
  The Patient Activation Measure-13 (PAM-13) is a concise assessment tool designed to evaluate an individual's knowledge, skills, and confidence in managing their own healthcare. Comprising 13 items, this self-report questionnaire helps healthcare professionals and researchers gauge a patient's level of activation and engagement in their healthcare journey. Respondents answer a series of questions related to their health-related knowledge, confidence in managing their health, and their proactivity in seeking healthcare information and making informed decisions. The score range from 13 to 52. Higher PAM-13 scores indicate a higher level of patient activation, which is often associated with better health outcomes and more effective self-management of chronic conditions.
Fatigue Severity | Baseline, hospital discharge, 1 month, 3 months and 6 months
  The perceived pain and Fatigue are measured with a Visual Analogue Scale from 0 to10, where 0 indicate no presence of pain or fatigue, and 10 indicate worst fatigue or pain.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, Chair, Study Director — Universidad de Granada
Locations (1):
- Faculty of Health Sciences. University of Granada., Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No